CLINICAL TRIAL: NCT05649670
Title: Prehospital Initiation of Reperfusion Therapy for Acute Ischemic Stroke: Randomized Medico-economic Evaluation of a Mobile Stroke Unit.
Brief Title: Acute Stroke: Prehospital Versus In-HospitAL Initiation of Recanalization Therapy- ASPHALT
Acronym: ASPHALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A02567-48; PRME 15-0677 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Acute
Keywords: Mobile Stroke Unit; MSU; Intravenous thrombolysis; Emergency Medical Service; Mechanical thrombectomy; Cost-utility; Cost-effectiveness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, PROBE design
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of 3-month mRS (via telephone interview)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (MSU) (Experimental): Deployment of MSU + conventional ambulance
  Interventions: Other: Mobile Stroke Unit deployment
- Control (usual care) (No Intervention): Deployment of conventional ambulance

INTERVENTIONS:
Other: Mobile Stroke Unit deployment — Deployment of an MSU + conventional ambulance, allowing prehospital CT-scan imaging with intracranial CT angiography. This will allow prehospital intravenous thrombolysis and optimal triage (i.e. accurate identification of patients with large vessel occlusion, who are eligible for mechanical thrombectomy).
  Other Names: Mobile Stroke Unit management
  Arms: Intervention (MSU)

SUMMARY:
ASPHALT is an academic-driven open-label randomized controlled trial of Mobile Stroke Unit (MSU) deployment versus standard care in France, with blinded assessment of efficacy endpoints. 450 patients with confirmed acute ischemic stroke will be recruited over a 3-year period, with 3-month follow-up.

DETAILED DESCRIPTION:
Instead of the traditional approach of waiting until the patient arrives at the hospital to perform brain imaging and start reperfusion therapies, mobile stroke units (MSUs; ambulances equipped with a CT scanner) now allow pre-hospital initiation of intravenous thrombolysis (IVT). Two large non-randomized clinical trials (B_PROUD & BEST-MSU) have recently shown that MSU use leads to improved functional outcomes at 3 months in specific settings. However, MSUs have been criticized because of their cost and a lack of evidence of a significant reduction in the time between symptom onset and mechanical thrombectomy, which is the cornerstone of treatment of patients with large vessel occlusion.

We hypothesized that compared to usual care, the deployment of a MSU would result in an incremental cost-utility ratio ≤50,000 euros per QALY in the lifetime horizon, even in an area with many thrombectomy-capable centers..

Academic-driven open-label randomized controlled trial of Mobile Stroke Unit (MSU) deployment versus standard care in France, with blinded assessment of efficacy endpoints. Randomization will be performed on an individual patient basis (randomization of MSU deployment at dispatch). 450 patients with confirmed acute ischemic stroke (emergency call ≤6 hours after onset) will be recruited over a 3-year period, with 3-month follow-up. Costs and clinical outcomes will be collected prospectively during the study period and used to extrapolate the incremental cost-utility ratio over a lifetime horizon.

ELIGIBILITY:
Inclusion Criteria:

* Emergency call to one of the two following emergency medical service (EMS) dispatch centers : SAMU (Service d'Aide Médicale Urgente) or BSPP (Brigade des Sapeurs Pompiers de Paris), between 08:00 and 18:00, 5 days a week (Monday to Friday).
* Suspected acute stroke according to a dispatcher stroke identification algorithm, adapted from the ROSIER scale
* Symptom onset-to-randomization time ≤ 6h
* Patient located within the predefined catchment area of the MSU
* MSU available at the time of the EMS call
* Informed consent (as approved by the ethics committee, informed consent will be obtained after randomization: at the arrival of the MSU (intervention group), or at hospital arrival (control group))

Exclusion Criteria:

* Patient confined to be more than 50% of waking hours
* Unknown or uncertain onset time (e.g. wake-up stroke)
* Medical history of epilepsy
* Recent epileptic seizure (<12 hrs)
* Suspicion of pregnancy
* Parturient or breastfeeding woman
* Patient already participating in another interventional study, which could influence the mRS at 3 months.
* Patient under guardianship or curatorship
* Patient not affiliated to French Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Utility Ratio (ICUR) | 3 months
  ICUR in the lifetime horizon, based on extrapolated results of the Modified Rankin Scale (mRS) at 3 months and incremental costs prospectively collected during the first 3 months
Key secondary outcome: Modified Rankin Scale (mRS) at 3 months | 90 +/- 14 days
  Modified Rankin scale, assessed in a blinded fashion (range, 0 to 6, with 0 indicating no disability, 3 indicating moderate disability, and 6 indicating death)

SECONDARY OUTCOMES:
ICUR at 3 months | 90 +/- 14 days
  Incremental Cost-Utility Ratio based on results of the Modified Rankin Scale (mRS) at 3 months and incremental costs prospectively collected during the first 3 months
ICUR at 5 years | 5 years
  Incremental Cost-Utility Ratio based on extrapolated results of the Modified Rankin Scale (mRS) at 3 months and incremental costs prospectively collected during the first 3 months
Time from symptom onset to intravenous thrombolysis (IVT) | up to 4.5 hours from symptom onset
  Time from symptom onset to IVT bolus
Time from symptom onset to mechanical thrombectomy (MT) | up to 24 hours from symptom onset
  Time from symptom onset to arterial puncture
Time from alarm to IVT | up to 4.5 hours from symptom onset
  Time from ambulance dispatch to IVT bolus
Time from alarm to MT | up to 24 hours from symptom onset
  Time from ambulance dispatch to arterial puncture
Death within 3 months after randomization | Within 90 days after randomization
  All-cause mortality
Death within 7 days after randomization | Within 7 days after randomization
  All-cause mortality
Proportion of ischemic stroke patients treated with IVT | up to 4.5 hours from symptom onset
  Proportion of patient treated with IVT among those with confirmed ischemic stroke
Proportion of ischemic stroke patients with MT | up to 24 hours from symptom onset
  Proportion of patient treated with MT among those with confirmed ischemic stroke
Proportion of ischemic stroke patients treated with IVT within 60 minutes of symptom onset | within 60 minutes of symptom onset
  Golden hour thrombolysis
Symptomatic intracranial hemorrhage | Within 36 hours from randomization
  ECASS-2 definition

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume TURC, MD, PhD, Principal Investigator — GHU Paris Psychiatrie et Neurosciences; Benoît VIVIEN, MD, PhD, Study Director — APHP - Centre Hospitalier Universitaire Necker
Locations (11):
- France (11):
  - AP-HP - hôpital Raymond Poincaré, Garches
  - AP-HP - hôpital Bicêtre, Le Kremlin-Bicêtre
  - AP-HP - hôpital Lariboisière, Paris
  - AP-HP - hôpital de la Pitié-Salpêtrière, Paris
  - GHU Paris psychiatrie & neurosciences, Paris
  - SAMU 75 de Paris, Paris
  - BSPP, Brigade des Sapeurs-Pompiers de Paris, Paris
  - AP-HP - hôpital Bichat - Claude-Bernard, Paris
  - Fondation Ophtalmologique Rothschild, Paris
  - Hôpital Saint Joseph, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) could be available to other researcher aiming to conduct an IPD-meta analysis of studies of MSU vs. usual care (please see access criteria below).
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Data sharing must respect the agreements made with funders. Teams wishing to obtain IPD must meet the sponsor and PI team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and time frame. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Turc G, Hadziahmetovic M, Walter S, Churilov L, Larsen K, Grotta JC, Yamal JM, Bowry R, Katsanos AH, Zhao H, Donnan G, Davis SM, Hussain MS, Uchino K, Helwig SA, Johns H, Weber JE, Nolte CH, Kunz A, Steiner T, Sacco S, Ebinger M, Tsivgoulis G, Fassbender K, Audebert HJ. Comparison of Mobile Stroke Unit With Usual Care for Acute Ischemic Stroke Management: A Systematic Review and Meta-analysis. JAMA Neurol. 2022 Mar 1;79(3):281-290. doi: 10.1001/jamaneurol.2021.5321. PMID 35129584